CLINICAL TRIAL: NCT00227682
Title: A Phase II Study of Arsenic Trioxide in Combination With Thalidomide, Dexamethasone, and Ascorbic Acid
Brief Title: Arsenic Trioxide, Thalidomide, Dexamethasone, and Ascorbic Acid in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated early due to funding suspension by grant sponsor.
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000443708; OHSU-1277 (Other: OHSU IRB); OHSU-HEM-03100-L (Other: OHSU Knight Cancer Institute); P30CA069533 (NIH)
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2010-06

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Ascorbic Acid; Arsenic Trioxide; Dexamethasone; Thalidomide

ARMS (1):
- Arsenic Trioxide (Experimental): Arsenic Trioxide in Combination With Thalidomide, Dexamethasone, and Ascorbic Acid
  Interventions: Dietary Supplement: ascorbic acid; Drug: arsenic trioxide; Drug: dexamethasone; Drug: thalidomide

INTERVENTIONS:
Dietary Supplement: ascorbic acid
Drug: arsenic trioxide
Drug: dexamethasone
Drug: thalidomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as arsenic trioxide, dexamethasone, and ascorbic acid, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells. Sometimes when chemotherapy is given, it does not stop the growth of cancer cells. The cancer is said to be resistant to chemotherapy. Giving arsenic trioxide together with chemotherapy may reduce drug resistance and allow the cancer cells to be killed. Thalidomide may stop the growth of multiple myeloma by blocking blood flow to the cancer. Giving arsenic trioxide together with thalidomide, dexamethasone, and ascorbic acid may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving arsenic trioxide together with thalidomide, dexamethasone, and ascorbic acid works in treating patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and side effects of arsenic trioxide administered in combination with thalidomide, dexamethasone, and ascorbic acid in patients with relapsed or refractory multiple myeloma.
* Determine, preliminarily, the anticancer effects of this regimen in these patients.
* Determine the duration of anticancer effects in patients treated with this regimen.
* Determine the effect of this regimen on bone and immune function in these patients.

OUTLINE: Patients receive arsenic trioxide IV continuously and oral ascorbic acid once daily on days 1-5 in week 1 and twice weekly in weeks 2-12 and oral thalidomide once daily in weeks 1-14. Treatment with arsenic trioxide, ascorbic acid, and thalidomide repeats every 14 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity. Patients also receive oral dexamethasone once daily on days 1-4. Treatment with dexamethasone repeats every 28 days.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma (MM)

  * Relapsed or refractory disease
* Monoclonal immunoglobulin spike by serum electrophoresis of ≥ 1 gm/dL AND/OR urine monoclonal immunoglobulin spike of ≥ 200 mg/24 hours
* Has received ≥ 2 prior treatment regimens for MM
* None of the following are allowed:

  * Non-secretory MM
  * Plasma cell leukemia
  * Polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-2

Life expectancy

* More than 3 months

Hematopoietic

* Platelet count ≥ 50,000/mm^3 (30,000/mm^3 if the bone marrow is extensively infiltrated)
* Hemoglobin ≥ 8.0 g/dL
* Absolute neutrophil count ≥ 1,000/mm^3

Hepatic

* AST and ALT < 3.0 times upper limit of normal (ULN)
* Bilirubin < 2.0 times ULN

Renal

* Not specified

Cardiovascular

* No cardiac disease, including any of the following conditions:

  * History of recurrent supraventricular arrhythmia
  * History of sustained ventricular tachycardia
  * History of second or third degree AV block
  * History of left bundle branch block
  * Cardiomyopathy with LVEF < 40%
  * Uncontrolled ischemic heart disease
* No myocardial infarction within the past 6 months
* No prolonged QT interval > 500 ms

Other

* Not pregnant or nursing
* Negative pregnancy test
* No HIV positivity
* No neuropathy > grade 3
* Potassium ≥ 4 mEq/L
* Magnesium ≥ 1.8 mg/dL

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* More than 30 days since prior investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2004-06; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Response rate (complete response, partial response, and minimal response) as measured by bone marrow aspirate, biopsy, cytogenetic analysis, serum, urine, and immunofixation skeletal survey at 6 months and end of study treatment

SECONDARY OUTCOMES:
Safety and tolerability as measured by physical exams, blood tests, and adverse events reports weekly

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Simic, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States